CLINICAL TRIAL: NCT03190213
Title: Pembrolizumab for the Treatment of Recurrent High Grade Neuroendocrine Carcinoma
Acronym: Pembro NEC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Update on clinical development: after discussions with the drug manufacturer, the PI has decided to discontinue the trial.
Sponsor: University of Utah (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI102310
Record Dates: First submitted 2017-06-13; First posted 2017-06-16 (Actual); Results first posted 2020-01-27 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Neuroendocrine Tumors
Keywords: high grade
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is an open label, non-randomized phase 2 study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab, all patients (Experimental)
  Interventions: Drug: Pembrolizumab Injection

INTERVENTIONS:
Drug: Pembrolizumab Injection — Pembrolizumab at a dose of 200 mg will be administered as an IV infusion over 30 minutes every 3 weeks until disease recurrence or discontinuation due to unacceptable toxicity for a maximum of 2 years. We anticipate on average patients will remain on treatment for approximately 24 weeks.

SUMMARY:
This is an open label, non-randomized phase 2 study to assess overall response rate (ORR), clinical benefit rate (CBR), overall survival (OS) and progression free survival (PFS) in patients with high grade neuroendocrine tumors treated with pembrolizumab 200mg Q 3 Weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, metastatic or unresectable neuroendocrine carcinoma of non-pulmonary origin, high grade as indicated by Ki-67 >20% and/or > 20 mitoses/10 hpf. Patients must have existing Ki-67 results from archival tissue or available tissue for Ki-67 testing. If no archival tissue is available the subject must agree to a fresh biopsy for testing to qualify for the study.
* Patients must have progressed during or after first-line treatment for metastatic or unresectable disease with either a platinum-based regimen (e.g. carboplatin + etoposide (VP-16), cisplatin + VP-16, FOLFOX) OR temozolomide-based regimen. Patients must have failed at least one line of therapy but no maximum number of therapies is exclusionary (i.e. second-line therapy and beyond).
* Have measurable disease based on Immune-Related Response Evaluation Criteria in Solid Tumors (irRECIST).
* Be greater than or equal to 18 years of age on day of signing informed consent.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Demonstrate adequate organ function as defined in the protocol, all screening labs should be performed within 14 days of treatment initiation.
* Subjects with a history of known central nervous system (CNS) metastases must have documentation of stable or improved brain imaging for at least 2 weeks after completion of definitive treatment. Definitive treatment may include surgical resection, whole brain irradiation, and/or stereotactic radiation therapy.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Must have recovered from adverse effects of any prior surgery, radiotherapy or other antineoplastic therapy.
* Last dose of any antineoplastic therapy greater than or equal to 2 weeks (including chemotherapy, small molecule inhibitors, radiation, and/or other investigational anticancer agents). Patients receiving hormone manipulation (e.g. selective estrogen receptor modulators (SERMs), aromatase inhibitors, luteinizing hormone-releasing hormone (LHRH} agonist, etc.) for reasons other than treatment of metastatic breast cancer may continue this treatment at the discretion of the investigator.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 2 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or receiving steroid therapy of any other form of immunosuppressive therapy within 7 days prior to first dose of trial treatment. Subjects who receive daily steroid replacement therapy serve as an exception to this rule. Daily prednisone at doses of 5 to 7.5 mg (or hydrocortisone equivalent doses) is an example of replacement therapy.
* Has a known history of active Bacillus Tuberculosis (TB).
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., less than or equal to Grade 1 or at baseline) from adverse events due to a previously administered agent. Note: Subjects with less than or equal to Grade 2 neuropathy are an exception to this criterion and may qualify for the study. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy. Patients receiving hormone manipulation (e.g. tamoxifen, aromatase inhibitors, LHRH agonist, etc.) for reasons other than treatment of metastatic breast cancer may continue this treatment at the discretion of the investigator.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer. Patients on long-term adjuvant therapy with no evidence of disease are not excluded if felt appropriate by investigator.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 2 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-programmed death (PD) -1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., hepatitis C virus (HCV) RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2019-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab: All Patients: Pembrolizumab 200 mg will be administered as an IV infusion every 3 weeks.
Period: Overall Study
Arm/Group | Pembrolizumab: All Patients
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab: All Patients
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.17 (17.03)
Age, Continuous [Median (Full Range); unit: years] | 44 [34 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response was measured using Immune Related Response Evaluation Criteria in Solid Tumors (irRECIST). At baseline, lesions found on CT or MRI imaging are cataloged as "target" or "non-target" lesions, and the longest dimensions of target lesions (or shortest dimension of target lymph nodes) are summed. irRECIST defines Complete Response (irCR) as a complete disappearance of all lesions after baseline. Partial Response (irPR) is defined as a 30% or more decrease in the target lesion measurements. Overall response rate is defined the percentage of participants with a best response of irCR + irPR.
Time Frame: planned for up to two years from baseline; actual time was up to 230 days (average of 70.5 days)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab: All Patients
Number analyzed (Participants) | 6
percentage of participants | 0 [0 to 45.9]

2. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit was measured using irRECIST. At baseline, lesions found on CT or MRI imaging are cataloged as "target" or "non-target" lesions, and the longest dimensions of target lesions (or shortest dimension of target lymph nodes) are summed. irRECIST defines irCR as a complete disappearance of all lesions after baseline. irPR is defined as a 30% or more decrease in the target lesion measurements. Progressive Disease (irPD) is a defined as a 20% or more increase in target lesion measurements. Stable Disease (irSD) is neither a sufficient shrinkage to qualify as irPR or irCR nor an increase that would qualify as irPD. Clinical Benefit Rate is defined as the percentage of participants with a best response of irCR + irPR + irSD.
Time Frame: planned for up to two years from baseline; actual time was up to 230 days (average of 70.5 days)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab: All Patients
Number analyzed (Participants) | 6
percentage of participants | 16.7 [0.4 to 64.1]

3. Secondary Outcome: Median Progression Free Survival
Description: Progression free survival (PFS) is the length of time during and after treatment that a participant lives and the disease does not get worse. PFS was measured as the time from first dose of pembrolizumab until disease progression by irRECIST criteria (>= 20% increase in target lesion measurements), and is reported as the median number of days patients survived without disease progression as calculated by the Kaplan-Meier method.
Time Frame: planned for up to four years from baseline; actual time was up to 230 days (average of 70.5 days)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pembrolizumab: All Patients
Number analyzed (Participants) | 6
days | 42.5 [40 to NA] — Value is infinity because there were too few patients to get a number.

4. Secondary Outcome: Median Overall Survival
Description: Overall survival (OS) is the length of time from the start of treatment that a participant lives. OS was measured as the time from first dose of pembrolizumab until the death of the participant or the end of follow-up (whichever was first), and is reported as the median number of days patients survived as calculated by the Kaplan-Meier method. This study was intended to follow participants up to four years after the initiation of study treatment, but the study and the follow-up period were terminated prematurely. The maximum follow up was 360 days.
Time Frame: planned for up to four years from baseline; actual time was up to 230 days (average of 70.5 days)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pembrolizumab: All Patients
Number analyzed (Participants) | 6
days | 262 [108 to NA] — Value is infinity because there were too few patients to get a number.

5. Secondary Outcome: Number of Patients With Adverse Events Reported
Description: Adverse Events were reported using the Common Terminology Criteria for Adverse Events (CTCAE) version 4. Each adverse event reported is assigned a severity grade from 1 to 5, where 1 is mild, 2 is moderate, 3 is severe, 4 is life threatening, and 5 indicates the event resulted in death. The number of patients experiencing any Grade 1-2 event and the number of patients experiencing any Grade 3 event are reported. There were no Grade 4 or Grade 5 events reported on this study. AEs were reported during study treatment and up to 90 days after last dose of treatment.
Time Frame: planned for up to two years of treatment plus 90 days; actual time was up to 338 days (average of 170 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab: All Patients
Number analyzed (Participants) | 6
Participants
  Grade 1-2 Event | 5
  Grade 3 Event | 5

ADVERSE EVENTS:
Time Frame: from the first dose of pembrolizumab until 30 days (for other adverse events) or 90 days (for serious adverse events) after last dose of pembrolizumab (average duration of 170 days, max duration of 338 days)
Description: The occurrence of adverse events was sought by non-directive questioning of the patient at each visit or phone contact during the study. Adverse events were also detected when they were volunteered by the patient during or between visits or through physical examination, laboratory test, or other assessments.
Arm/Group | Pembrolizumab: All Patients
All-Cause Mortality (participants affected / at risk) | 2/6
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab: All Patients (N=6)
Abdominal pain (Gastrointestinal disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab: All Patients (N=6)
Abdominal pain (Gastrointestinal disorders) | 3
Allergic reaction (Immune system disorders) | 1
Anal pain (Gastrointestinal disorders) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (3)
Autoimmune disorder (Immune system disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 3 (4)
Headache (Nervous system disorders) | 1
Hot flashes (Vascular disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infections and infestations - Other: Thrush (Infections and infestations) | 1
Infusion related reaction (General disorders) | 1
Insomnia (Psychiatric disorders) | 1 (2)
Lymph node pain (Blood and lymphatic system disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Nausea (Gastrointestinal disorders) | 4
Nervous system disorders - Other: Allodynia (Nervous system disorders) | 1 (2)
Pain (General disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rectal pain (Gastrointestinal disorders) | 1
Restlessness (Psychiatric disorders) | 1
Seizure (Nervous system disorders) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Spasticity (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT03190213/Prot_SAP_000.pdf